CLINICAL TRIAL: NCT02489019
Title: Fentanyl Effect on Blood Pressure in Elderly Patients After Induction of General Anesthesia
Acronym: Fentanyl
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Jeffrey Hartwig, Assistant Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 204821
Record Dates: First submitted 2015-07-01; First posted 2015-07-02 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Hypotension
Keywords: Anesthesia; Fentanyl; Elderly
MeSH Terms: conditions — Hypotension | interventions — Sodium Chloride; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Placebo Comparator): Individuals assigned to this condition will receive 0.9 mcg/kg sodium chloride (NaCL)
  Interventions: Drug: Sodium chloride
- Low Dose (Experimental): Individuals assigned to this condition will receive 1 mcg/kg fentanyl
  Interventions: Drug: Fentanyl
- High Dose (Experimental): Individuals assigned to this condition will receive 2 mcg/kg fentanyl
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Sodium chloride — Sodium chloride will be used as a placebo comparator in this trial
  Other Names: NaCL
  Arms: Control
Drug: Fentanyl — Fentanyl is a synthetic opioid analgesic that will be used as the experimental intervention in this trial
  Other Names: Actiq; Duragesic; Fentora; Sublimaze
  Arms: High Dose; Low Dose

SUMMARY:
Hypotension is frequently encountered after induction of general anesthesia. It can be pronounced in elderly patients and can require administration of vasopressor agents including ephedrine and phenylephrine. Intraoperative hypotension, especially prolonged episodes, can contribute to an increase in morbidity and mortality in the postoperative period as suggested by some former studies. The investigators hypothesize that fentanyl can contribute to the decrease in blood pressure (BP) that is seen after induction of general anesthesia in older patients. This hypotension may be due to fentanyl blocking effect on the sympathetic nervous system.

This study will be the first one to examine the effect of fentanyl administration on blood pressure in elderly patients with induction of general anesthesia prior to the start of surgery. If the study shows that fentanyl contributes to hypotension during this period, it may lead to a change in practice and better patient outcomes and mortality rates.

DETAILED DESCRIPTION:
This is a prospective double-blinded randomized controlled trial (RCT) where patients will be assigned randomly by the investigational pharmacist. Patients will be assigned to one of three groups: (1) A control group that receives 0.9 mcg/kg sodium chloride (NaCL), (2) a fentanyl group that receives 1 mcg/kg fentanyl, or (3) a fentanyl group that receives 2 mcg/kg fentanyl.

The definition of intraoperative hypotension in this study is defined as a mean blood pressure (MAP) less than 25% compared to the baseline value (i.e., the participants' first blood pressure reading after entering the operating room). All study drug agents will be dispensed by the pharmacy in five milliliter syringes labeled as "study medication". The volume of any of the three study medication will be adjusted by the pharmacist to reflect an equal volume.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60 years and older
* Patients coming from home (including those who will be admitted post-operatively)
* Surgeries with general anesthesia alone or if combined with peripheral nerve blocks
* Patients must be seen at the Russo operating room at Loyola Medical Center (Maywood, IL)

Exclusion Criteria:

* Age less than 60
* Patient refusal
* Inpatient or emergency cases
* Patients having combined general anesthesia and epidural anesthesia
* Patients with a pre-induction mean arterial blood pressure (MAP) less than 50 or greater than 150
* Patients who will receive rapid sequence induction with succinylcholine
* Patients scheduled for cardiovascular surgery
* Patients scheduled for inhalational induction
* Patients with weight greater than 125 kg
* Patients with a history of chronic opioid use

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2018-02-19 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Development of hypotension | At 60 minutes following dose administration
  Blood pressure will be recorded 60 minutes after administration of the study agent

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Hartwig, MD, Principal Investigator — Loyola University Chicago
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bijker JB, van Klei WA, Vergouwe Y, Eleveld DJ, van Wolfswinkel L, Moons KG, Kalkman CJ. Intraoperative hypotension and 1-year mortality after noncardiac surgery. Anesthesiology. 2009 Dec;111(6):1217-26. doi: 10.1097/ALN.0b013e3181c14930. PMID 19934864
- [Background] Bijker JB, van Klei WA, Kappen TH, van Wolfswinkel L, Moons KG, Kalkman CJ. Incidence of intraoperative hypotension as a function of the chosen definition: literature definitions applied to a retrospective cohort using automated data collection. Anesthesiology. 2007 Aug;107(2):213-20. doi: 10.1097/01.anes.0000270724.40897.8e. PMID 17667564
- [Background] Billard V, Moulla F, Bourgain JL, Megnigbeto A, Stanski DR. Hemodynamic response to induction and intubation. Propofol/fentanyl interaction. Anesthesiology. 1994 Dec;81(6):1384-93. doi: 10.1097/00000542-199412000-00013. PMID 7992907
- [Background] Reich DL, Hossain S, Krol M, Baez B, Patel P, Bernstein A, Bodian CA. Predictors of hypotension after induction of general anesthesia. Anesth Analg. 2005 Sep;101(3):622-628. doi: 10.1213/01.ANE.0000175214.38450.91. PMID 16115962
- [Background] Monk TG, Saini V, Weldon BC, Sigl JC. Anesthetic management and one-year mortality after noncardiac surgery. Anesth Analg. 2005 Jan;100(1):4-10. doi: 10.1213/01.ANE.0000147519.82841.5E. PMID 15616043